CLINICAL TRIAL: NCT01481935
Title: Use of an Enhanced Room Cleaning Protocol in the Intensive Care Unit to Reduce Contamination of Disposable Isolation Gowns and Gloves With Methicillin-resistant Staphylococcus Aureus and Multi-drug Resistant Acinetobacter Baumannii
Brief Title: Enhanced Room Cleaning in Intensive Care Units to Reduce Gown and Glove Contamination With Multi-drug-resistant Bacteria
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Anthony Harris, Professor, Department of Epidemiology and Public Health, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: HP-00048554
Record Dates: First submitted 2011-11-21; First posted 2011-11-30 (Estimated); Results first posted 2012-10-19 (Estimated); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Infection Control
Keywords: Antibiotic resistant bacteria; Colonization; Hospital cleaning; Environmental cleaning; Infection Control

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Enhanced Cleaning (Experimental): Rooms in the Enhanced Cleaning arm will receive cleaning of frequently contaminated surfaces by a study researcher in addition to standard room cleaning by hospital housekeeping staff.
  Interventions: Other: Enhanced cleaning of surfaces in ICU rooms
- Sham Enhanced Cleaning (Sham Comparator): Rooms in the Sham Enhanced Cleaning arm will receive a sham cleaning of frequently contaminated surfaces by a study researcher in addition to standard room cleaning by hospital housekeeping staff.
  Interventions: Other: Sham enhanced cleaning of surfaces in ICU rooms

INTERVENTIONS:
Other: Enhanced cleaning of surfaces in ICU rooms — Using a paper towel pre-soaked with a commercially-available quaternary ammonium cleaning solution (Virex WetTask wipes, Kimberly-Clark, Irving, Texas), the following surfaces will be wiped clean by a study investigator if present: bed rail top bar, bed electronic control surfaces, moveable tray table top and control surfaces desktop and sides, IV poles, infusion pump control surfaces, nurse call button, patient telephone/remote control, sink console top, light switches and plates, supply cart top and drawer handles, ventilator control surfaces and desk, vital signs monitor control surfaces. Cleaning will occur once on the day of enrollment and follow-up.
  Other Names: Environmental cleaning
  Arms: Enhanced Cleaning
Other: Sham enhanced cleaning of surfaces in ICU rooms — While holding a paper towel pre-soaked with a commercially-available quaternary ammonium cleaning solution (Virex WetTask wipes, Kimberly-Clark, Irving, Texas), a study investigator will mime the action of wiping the following surfaces in the room clean if present: bed rail top bar, bed electronic control surfaces, moveable tray table top and control surfaces desktop and sides, IV poles, infusion pump control surfaces, nurse call button, patient telephone/remote control, sink console top, light switches and plates, supply cart top and drawer handles, ventilator control surfaces and desk, vital signs monitor control surfaces. The sham cleaning will occur once on the day of enrollment and follow-up.
  Other Names: Sham Environmental Cleaning
  Arms: Sham Enhanced Cleaning

SUMMARY:
The purpose of this study is to determine whether extra cleaning of frequently-contaminated surfaces in intensive care rooms is effective in preventing contamination of disposable isolation gowns and gloves with multi-drug resistant bacteria.

DETAILED DESCRIPTION:
Hospital infections are often caused by bacteria such as methicillin-resistant Staphylococcus aureus (MRSA) or multi-drug-resistant Acinetobacter baumannii (MDRAB). Hospital infections increase the cost of health care, length of hospital stay, and mortality compared to infections with antibiotic-susceptible organisms. Many of these antibiotic-resistant bacteria are transmitted by patient-to-patient contact.

Healthcare workers are one possible vector of patient-to-patient transmission. Transient colonization of hands, clothing and protective equipment can leads to the colonization and infection of other patients. The surfaces of patient rooms are also frequently contaminated with antibiotic-resistant bacteria. A number of recent studies have concluded that patient rooms are not cleaned thoroughly or frequently enough to keep commonly touched surfaces free of bacterial contamination. Given the frequency of contact between the healthcare worker and the patient's environment, bacteria that contaminate environmental surfaces while the patient is in the room are a significant potential reservoir for patient-to-patient transmission via the hands of healthcare workers.

In this study, the investigators will examine rooms of intensive care unit patients colonized with MRSA or MDRAB. The investigators will randomize these rooms to receive either standard room cleaning plus a cleaning of high-touch surfaces ('enhanced cleaning') or to receive only standard room cleaning plus a sham cleaning of high-touch surfaces ('sham enhanced cleaning'). The investigators will then culture healthcare workers' disposable isolation gowns and gloves as they exit the enrolled room after routine patient care activities. The investigators will examine the cultures for the presence of MRSA or MDRAB to determine whether additional cleaning significantly reduces the proportion of healthcare workers with contaminated gloves and gowns, and therefore may reduce the risk of transmitting these bacteria to other patients. The results of this trial will help guide future efforts to decrease patient-to-patient transmission of antibiotic-resistant bacteria.

ELIGIBILITY:
Inclusion Criteria:

* Room is occupied by a patient colonized with methicillin-resistant Staphylococcus aureus and/or multi-drug-resistant Acinetobacter baumannii
* Occupant of the room is on contact precautions
* Occupant was admitted to the room at least 24 hours prior to the time of screening

Exclusion Criteria:

* Room is occupied by a patient who occupied another room at the time it was enrolled and followed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2011-08; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony D Harris, MD MPH, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- University of Maryland, Baltimore, Baltimore, Maryland, United States

REFERENCES:
- [Background] Carling PC, Von Beheren S, Kim P, Woods C; Healthcare Environmental Hygiene Study Group. Intensive care unit environmental cleaning: an evaluation in sixteen hospitals using a novel assessment tool. J Hosp Infect. 2008 Jan;68(1):39-44. doi: 10.1016/j.jhin.2007.09.015. Epub 2007 Dec 11. PMID 18069083
- [Background] Goodman ER, Platt R, Bass R, Onderdonk AB, Yokoe DS, Huang SS. Impact of an environmental cleaning intervention on the presence of methicillin-resistant Staphylococcus aureus and vancomycin-resistant enterococci on surfaces in intensive care unit rooms. Infect Control Hosp Epidemiol. 2008 Jul;29(7):593-9. doi: 10.1086/588566. PMID 18624666
- [Background] Morgan DJ, Liang SY, Smith CL, Johnson JK, Harris AD, Furuno JP, Thom KA, Snyder GM, Day HR, Perencevich EN. Frequent multidrug-resistant Acinetobacter baumannii contamination of gloves, gowns, and hands of healthcare workers. Infect Control Hosp Epidemiol. 2010 Jul;31(7):716-21. doi: 10.1086/653201. PMID 20486855
- [Background] Carling PC, Bartley JM. Evaluating hygienic cleaning in health care settings: what you do not know can harm your patients. Am J Infect Control. 2010 Jun;38(5 Suppl 1):S41-50. doi: 10.1016/j.ajic.2010.03.004. PMID 20569855
- [Background] Boyce JM, Potter-Bynoe G, Chenevert C, King T. Environmental contamination due to methicillin-resistant Staphylococcus aureus: possible infection control implications. Infect Control Hosp Epidemiol. 1997 Sep;18(9):622-7. PMID 9309433
- [Background] Snyder GM, Thom KA, Furuno JP, Perencevich EN, Roghmann MC, Strauss SM, Netzer G, Harris AD. Detection of methicillin-resistant Staphylococcus aureus and vancomycin-resistant enterococci on the gowns and gloves of healthcare workers. Infect Control Hosp Epidemiol. 2008 Jul;29(7):583-9. doi: 10.1086/588701. PMID 18549314
- [Background] Wilson AP, Smyth D, Moore G, Singleton J, Jackson R, Gant V, Jeanes A, Shaw S, James E, Cooper B, Kafatos G, Cookson B, Singer M, Bellingan G. The impact of enhanced cleaning within the intensive care unit on contamination of the near-patient environment with hospital pathogens: a randomized crossover study in critical care units in two hospitals. Crit Care Med. 2011 Apr;39(4):651-8. doi: 10.1097/CCM.0b013e318206bc66. PMID 21242793
- [Derived] Hess AS, Shardell M, Johnson JK, Thom KA, Roghmann MC, Netzer G, Amr S, Morgan DJ, Harris AD. A randomized controlled trial of enhanced cleaning to reduce contamination of healthcare worker gowns and gloves with multidrug-resistant bacteria. Infect Control Hosp Epidemiol. 2013 May;34(5):487-93. doi: 10.1086/670205. PMID 23571365

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Rooms in 4 ICUs in a large, urban, academic hospital. Recruitment began on 7/21/2011 and ended on 5/20/2012.
Groups:
- Sham Enhanced Cleaning: Rooms in the Sham Enhanced Cleaning arm received a single sham extra cleaning of frequently contaminated surfaces by a study researcher in addition to standard room cleaning by hospital housekeeping staff. Sham Enhanced Cleaning was performed once per day of enrollment and follow-up. Seventeen surfaces identified by the CDC as being 'frequently touched and frequently contaminated' were cleaned as part of the experimental intervention. Cleaning was performed using standard hospital cleaning products (wipes soaked in a commercially-available quaternary ammonium solution).
- Enhanced Cleaning: Rooms in the Enhanced Cleaning arm received a single extra cleaning of frequently contaminated surfaces by a study researcher in addition to standard room cleaning by hospital housekeeping staff. Enhanced Cleaning was performed once per day of enrollment and follow-up. Seventeen surfaces identified by the CDC as being 'frequently touched and frequently contaminated' were cleaned as part of the experimental intervention. Cleaning was performed using standard hospital cleaning products (wipes soaked in a commercially-available quaternary ammonium solution).
Period: Overall Study
Arm/Group | Sham Enhanced Cleaning | Enhanced Cleaning
Started | 97 | 93
Completed | 97 | 93
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Enhanced Cleaning | Sham Enhanced Cleaning | Total
Number analyzed (Participants) | 93 | 97 | 190
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 66 | 66 | 132
  >=65 years | 27 | 31 | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 51 (19) | 56 (17) | 54 (18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 41 | 71
  Male | 63 | 56 | 119
Region of Enrollment [Number; unit: participants]
  United States | 93 | 97 | 190

OUTCOME MEASURES:

1. Primary Outcome: Contamination of Disposable Isolation Gown and Gloves With Methicillin-resistant Staphylococcus Aureus or Multi-drug-resistant Acinetobacter Baumannii
Description: Swabs will be collected from the disposable gown and gloves of healthcare workers exiting the enrolled room. A single swab will be used for both gloves and the gown. The swab will be assayed for methicillin-resistant Staphylococcus aureus, multi-drug-resistant Acinetobacter baumannii, or both, depending on which organism(s) the occupant of the enrolled room is colonized with. The swab will be considered positive if the relevant organism is isolated. We will sample the first 15 healthcare worker exits after the room has received the allocated intervention.
Time Frame: As a healthcare worker exits the enrolled room (1 day)
Population: Unit of analysis was the ICU room. Results from multiple participants who occupied a single room over the course of the trial were summarized by room.
Measure: Mean (Standard Error); unit: percentage of positive cultures
Units Other Than Participants: Rooms
Arm/Group | Sham Enhanced Cleaning | Enhanced Cleaning
Number analyzed (Participants) | 97 | 93
Number analyzed (Rooms) | 55 | 49
percentage of positive cultures | 20.5 (2.1) | 17.2 (2.5)

ADVERSE EVENTS:
Arm/Group | Sham Enhanced Cleaning | Enhanced Cleaning
Serious Adverse Events (participants affected / at risk) | 0/97 | 0/93
Other Adverse Events (participants affected / at risk) | 0/97 | 0/93

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No